CLINICAL TRIAL: NCT02521129
Title: A New Track Ablation Device for Liver Biopsy: A Feasibility Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyunchul Rhim, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-11-048-003; GFO1130071 (Other Grant/Funding Number: Samsung Medical Center)
Record Dates: First submitted 2015-08-03; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ablation (Experimental): Intervention: ablation of biopsy needle track with a new device
  Interventions: Device: Biopsy Track Ablator (STARmed, Goyang, Korea)

INTERVENTIONS:
Device: Biopsy Track Ablator (STARmed, Goyang, Korea) — After percutaneous ultrasound guided biopsy for hepatic masses is performed, biopsy track is ablated with a new track ablation device.
  Other Names: Ultrasound (Logig E9, GE Healthcare)

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of a new biopsy track ablation device for liver biopsy.

DETAILED DESCRIPTION:
Background:

* Percutaneous biopsy for hepatic masses has a potential risk of bleeding and peritoneal tumor seeding.
* A new device for biopsy track ablation has been invented to reduce the risk of bleeding and peritoneal tumor seeding.

Method:

* Routine percutaneous biopsy for hepatic masses is performed.
* Immediate after obtaining tissue, biopsy needle track is ablated with a new biopsy tract ablator.
* Immediate (with ultrasound) and 24 hours (with CT scan) after procedure, occurrence of complications is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with a hepatic mass on CT scan or MRI
* patients who are referred for percutaneous biopsy of a hepatic mass
* patients with normal range of platelet count and coagulation test

Exclusion Criteria:

* pregnant women
* patients with ascites
* Uncooperative patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complications | within 24 hours after procedure
  If procedure-related complications are suspected clinically, appropriate tests such as CT scan or Ultrasound are performed and complications are evaluated.
  If procedure-related complications are not suspected, non-contrast CT scan is performed at 24 hours after procedure and complications are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hyunchul Rhim, professor, Principal Investigator — Samsung Medical Center

REFERENCES:
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666